CLINICAL TRIAL: NCT06456060
Title: Exploring the Efficacy of Pure Honey Dressing in Contrast to Alvogyl in the Resolution of Dry Socket: A Comparative Analysis
Brief Title: Efficacy of Pure Honey Dressing in Contrast to Alvogyl in the Resolution of Dry Socket
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Watim Medical & Dental College (Other)
Responsible Party: Principal Investigator, Muhammad Ilyas, Assistant Professor, Watim Medical & Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 639/NID/24
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Dry Socket
MeSH Terms: conditions — Dry Socket | interventions — butyl aminobenzoate, eugenol, iodoform, spearmint oil drug combinations; Honey

STUDY DESIGN:
Intervention Model Description: Patients will be divided into the following two groups:
  1. Study group
  2. Control group
  In the study group, after flushing the socket with normal saline, 2 ml of Honey soaked in a sterile gauze will be applied to cover the socket, whereas in the control group, a gauze with Alveogyl will be used to cover the socket instead of Honey.
Who Masked: Participant
Masking Description: Participants will be blinded about the use of honey or Alveogyl in the dressing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Alvogyl) Group (Active Comparator): In Control Group, after flushing the socket with normal saline a gauze soaked with Alvogyl will be used to cover the socket..
  Interventions: Drug: Alvogyl
- Study (Honey) Group (Experimental): In the Study (Honey) Group, after flushing the socket with normal saline, 2 ml of Honey soaked in a sterile gauze will be applied to cover the socket.
  Interventions: Drug: Honey

INTERVENTIONS:
Drug: Alvogyl — Alvogyl soaked in a sterile gauze will be applied to cover the socket.
  Arms: Control (Alvogyl) Group
Drug: Honey — Honey soaked in a sterile gauze will be applied to cover the socket.
  Arms: Study (Honey) Group

SUMMARY:
Dry socket, or Alveolar Osteitis, is the most common complication that can follow a tooth extraction. Over the years, various approaches have been employed to expedite the healing process and alleviate the associated symptoms. Among these, Alvogyl has been the most commonly used dry socket dressing all over the globe. However due to Alvogyl's potential side effect of causing a foreign body reaction & ultimately necrosis of the alveolar bone if left in the socket along with its high cost, scientists have sought to develop new techniques. Among them, Honey dressing has heralded promising properties in facilitating the resolution of dry socket, thus opening the window of a side-effect free natural viable alternative to Alvogyl. In this research, we aim to compare the efficacy of pure Honey as a dry socket dressing in comparison to Alvogyl.

DETAILED DESCRIPTION:
This will be an interventional study, carried out using a quasi-experimental design.

After making the diagnosis of Alveolar osteitis by means of clinical examination and radiograph, Demographic data along with other associated information such as their medical condition, tooth indicated for extraction, pre-operative pain, and halitosis will be documented.

With 20 patients in each, Patients will be divided into the following two groups:

1. Study group
2. Control group

In the study group, after flushing the socket with normal saline, 2 ml of Honey soaked in a sterile gauze will be applied to cover the socket, whereas in the control group, a gauze with Alveogyl will be used to cover the socket instead of Honey.

Patients will be allowed to continue their oral analgesic medication, namely Ibuprofen 200 mg, 400 mg, or 600 mg twice daily, depending upon the severity of initial pain upon diagnosis. Pain relief will be recorded and compared between the two groups on a visual analog pain scale at every appointment.

The intra-alveolar packing will be continued & will be kept being changed at regular intervals until the postoperative pain symptoms subside. Patients will be reviewed at 5 min post-medication, 30 min post-medication, 60 min post-medication, 2nd day post-medication, 4th day post-medication and 7th day post-medication. The patients will be requested to note daily pain records on a (0-10) visual analog scale, with 0 representing no pain and 10 representing the worst pain.

For safety purposes, any harmful effects of the medications will also be recorded. Patients will be instructed to call the investigator immediately about any problem & in such circumstances, treatment will be immediately terminated and discontinued. The patient will be requested to visit the investigator at the earliest possible time. If no side effects are noted, the treatment option will be repeated a maximum of four times over two weeks to assess the complete effect of the medication in case complete relief was not achieved the first time. The total time required for complete healing and the number of repeated sessions for each medication until complete relief from all symptoms will be recorded in Performa, attached as Annexure.

The success rate of the procedure will be categorized into excellent, good, fair, and poor, according to pain relief, the need to use oral analgesics and the number of repeated sessions for each medication.

Excellent: complete relief of pain without the use of analgesics; pain score = 0 (no pain) Good: complete relief of pain with modest use of analgesics (200 mg ibuprofen); pain score: 1-3 (mild) Fair: complete relief of pain with moderate use of analgesics (400 mg ibuprofen); pain score: 4-6 (moderate pain) Poor: continued pain despite high dose of analgesics (600 mg ibuprofen); pain score 7-10 (severe pain)

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age of both genders.
2. Patients who underwent extraction of teeth and were clinically diagnosed with dry socket at the OMFS department of NID, Multan.
3. Patients which give informed consent.

Exclusion Criteria:

1. Patients below the age of 18 and above the age of 70.
2. Patients with various bone diseases, including osteoporosis & a history of taking oral or intravenous bisphosphonates
3. Patients with a history of radiotherapy on the head, neck, and jawbones were excluded from this study,
4. Patients with systemic diseases such as diabetes mellitus, hepatic dysfunctions, blood dyscrasias, and bleeding disorders
5. Patients with allergy to Ibuprofen & honey
6. Patients having symptoms similar to dry socket due to retained root pieces, oroantral communication, or any bony or soft tissue pathology by the help of a radiograph
7. Patients who did not give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain relief | Patients will be reviewed at 5 min post-medication, 30 min post-medication, 60 min post-medication, 2nd day post-medication, 4th day post-medication and 7th day post-medication.
  The patients will be requested to note daily pain records on a (0-10) visual analog scale, with 0 representing no pain and 10 representing the worst pain..

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ilyas, MBBS, FCPS, Study Director — Watim Medical & Dental College
Locations (1):
- Nishtar Institute of Dentistry, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Keshini MP, Shetty SK, Sundar S, Chandan SN, Manjula S. Assessment of Healing Using Alvogyl and Platelet Rich Fibrin in Patients with Dry Socket - An Evaluative Study. Ann Maxillofac Surg. 2020 Jul-Dec;10(2):320-324. doi: 10.4103/ams.ams_259_19. Epub 2020 Dec 23. PMID 33708574
- [Result] Abu-Mostafa N, Al-Daghamin S, Al-Anazi A, Al-Jumaah N, Alnesafi A. The influence of intra-alveolar application of honey versus Chlorhexidine rinse on the incidence of Alveolar Osteitis following molar teeth extraction. A randomized clinical parallel trial. J Clin Exp Dent. 2019 Oct 1;11(10):e871-e876. doi: 10.4317/jced.55743. eCollection 2019 Oct. PMID 31636855
- [Result] Soni N, Singh V, Mohammad S, Singh RK, Pal US, Singh R, Aggrwal J, Pal M. Effects of honey in the management of alveolar osteitis: A study. Natl J Maxillofac Surg. 2016 Jul-Dec;7(2):136-147. doi: 10.4103/0975-5950.201354. PMID 28356684